CLINICAL TRIAL: NCT05058443
Title: Denosumab Protects Bone Loss and Function in Patients With Osteoporotic Vertebral Compression Fracture After Percutaneous Vertebroplasty: a Randomized Placebo-controlled Clinical Trial
Brief Title: Denosumab and Osteoporotic Vertebral Compression Fracture
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenzhenPH spine
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteoporotic Vertebral Compression Fracture
Keywords: denosumab; vertebroplasty
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): Denosumab 60 mg were injected subcutaneously every 6 months (Q6M)
  Interventions: Drug: Denosumab 60 mg/ml [Prolia]
- Placebo (Placebo Comparator): Equal volume of saline (0.9%) as placebo were injected subcutaneously every 6 months (Q6M)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab 60 mg/ml [Prolia] — denosumab subcutaneously every 6 months (Q6M)
  Other Names: Denosumab
  Arms: Denosumab
Drug: Placebo — placebo subcutaneously every 6 months (Q6M)
  Other Names: equal volume of saline (0.9%)
  Arms: Placebo

SUMMARY:
This study aimed to investigate the effect of denosumab on bone mineral density(BMD), bone turnover markers(BTMs), functional status, secondary fracture rate, and adverse effects in osteoporotic vertebral compression fracture (OVCF) patients after vertebroplasty during a 12-month follow-up period.

DETAILED DESCRIPTION:
We performed a single-center, placebo-controlled, randomized clinical trial in the Department of Spinal Surgery located at the First Affiliated Hospital of Southern University of Science and Technology (Shenzhen People's Hospital). All patients underwent vertebroplasty and randomly received denosumab treatment or placebo control after surgery. The BMDs (lumbar, total hip, and femoral neck) and BTMs were assessed at baseline, 6, and 12 months post-operation. The visual analog scale (VAS) score for back pain, and function status questionnaires, including EuroQol five-dimension (EQ-5D), the Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31), and the Roland-Morris Disability Functioning Questionnaire (RMDQ),secondary fracture rate, and adverse effects in OVCF patients after vertebroplasty during a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 50 and 90 years old
* X-ray diagnosis of 1 or 2 segment vertebral compression fractures from T4 to L5
* Bone mineral density T value less than -1 via dual-energy X-ray
* A recent fracture history less than 6 weeks
* MRI show bone marrow edema of fractured vertebrae
* low back pain, local paravertebral tenderness

Exclusion Criteria:

* Must be able to have no intervertebral fissure
* Must be able to have no infection
* Must be able to have no malignancy
* Must be able to have no neurological dysfunction
* Must be able to have no previous use of anti-osteoporosis drugs
* Must be able to have no inability to perform magnetic resonance imaging
* Must be able to have no prior back open surgery
* Must be able to have no other established contraindications for elective surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Procollagen type 1 n-terminal propeptide (P1NP) | up to 12 months
  Bone formation marker, P1NP were determined at baseline, 6 and 12 months after surgery.
C-terminal cross-linked type 1 collagen terminal peptide (CTX) | up to 12 months
  Bone resorption marker, CTX were determined at baseline, 6 and 12 months after surgery
Lumbar bone mineral density(BMD) | up to 12 months
  Lumbar vertebral (L1 to L4, except the surgery segment) BMD were determined at baseline, 6 and 12 months via dual-energy X-ray.
Total hip BMD | up to 12 months
  Total hip BMD were determined at baseline, 6 and 12 months via dual-energy X-ray.
Femoral neck BMD | up to 12 months
  Femoral neck BMD were determined at baseline, 6 and 12 month via dual-energy X-ray
Visual analog scale (VAS) back | up to 12 months
  The VAS score for back pain were determined at baseline, 6 and 12 month. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain.

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is scored by 24 adding up the number of items checked "yes" on different low back pain-related daily activity disabilities. Total scores range from 0 to 24, with higher scores 24 indicating a higher level of disability related to low back pain and lowest 0 represents no back pain.
The QUALEFFO-31 Questionnaire | up to 12 month
  The Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31), which contains three domains including pain, physical function, and mental function. This scale is assessed on a scale of 0 to 100, with 0 indicating the highest QoL and 100 the lowest.
The EQ-5D Questionnaire | up to 12 month
  The EQ-5D questionnaire evaluates health status consisting five dimensions: mobility, self-care, performance of usual activities, pain or discomfort, and anxiety or depression. After conversion, the index was between 0 and 1.0 (minimum score: 0, indicating worst health state; full score:1.0, indicating full health).
Secondary fracture rate | up to 12 month
  Secondary fracture rate containing vertebral fracture and non-vertebral fracture was assessed at 12 month after surgery. The lowest score was 0, the highest score was 100%. The lower score 0 represents no secondary fracture.
Adverse events | up to 12 month
  The main adverse events including deep venous thrombosis, pneumonia, acute renal failure, pulmonary embolism, myocardial infarction, influenza, transfer to intensive care unit, joint pain, headache, nausea, osteonecrosis of the jaw, atypical femoral fracture and rash.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Xiao, Doctor, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang R, Qian X, Xuan Z, Xu Y, Chen Y, Gu H, Fu C. Health related quality of life and its impacts by chronic diseases in urban community population, Shanghai, China in 2015. Psychol Health Med. 2021 Sep;26(8):931-939. doi: 10.1080/13548506.2020.1856896. Epub 2020 Dec 11. PMID 33305593
- [Result] Zhou C, Li Q, Huang S, Fan L, Wang B, Dai J, Tang X. Validation of the simplified Chinese version of the quality of life questionnaire of the European foundation for osteoporosis (QUALEFFO-31). Eur Spine J. 2016 Jan;25(1):318-324. doi: 10.1007/s00586-015-4066-z. Epub 2015 Jun 14. PMID 26070551
- [Result] Stevens ML, Lin CC, Maher CG. The Roland Morris Disability Questionnaire. J Physiother. 2016 Apr;62(2):116. doi: 10.1016/j.jphys.2015.10.003. Epub 2015 Dec 11. No abstract available. PMID 26687949